CLINICAL TRIAL: NCT00938067
Title: American Indian and Alaska Native Health Disparities Staying Connected: Trauma Center to Tribal Community Linkage for Physically Injured American Indian Patients
Brief Title: Staying Connected: Trauma Center to Tribal Community Linkage for Physically Injured American Indian Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Douglas Zatzick, Professor, University of Washington
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 35970-C; P60 MD0005-07
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Injuries
Keywords: Injuries, Trauma
MeSH Terms: conditions — Wounds and Injuries; Accidental Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Staying Connected: Care Management (Experimental): The intervention combines case management, psychopharmacological and culturally appropriate and individually tailored trauma support activities with evidence-based treatments.A key feature is the provision of a continuous healing relationship by a care management treatment team.The care manager, informed by the Native healer interviews, will provide a culturally appropriate and ongoing helping relationship to each intervention patient in the weeks and months post-injury and will remain in close contact with the trauma survivor subject for 6 months.Together, the care manager and trauma survivor subject will work on a plan to readjust to daily activities. The care management team will also coordinate psychopharmacological interventions for PTSD and related co-morbidities with primary care and or other community providers.
  Interventions: Behavioral: Staying Connected

INTERVENTIONS:
Behavioral: Staying Connected — The overarching goal of the Staying Connected intervention is to establish a compassionate and culturally sensitive treatment trajectory that diminishes posttraumatic suffering by reducing symptomatic distress, improving functional recovery, and reducing the risk of injury recurrence. This trajectory begins with surgical treatment and extends through outpatient care and community rehabilitation. The collaborative care intervention fundamentally restructures the delivery of mental health care within trauma care systems by bringing together providers currently working independently to form an interdisciplinary mental health team. Team members work together and in a liaison capacity with other trauma center providers and community practitioners in order to bridge care across service delivery sectors.

SUMMARY:
The purpose of this study is to provide American Indian trauma patients, treated at the Harborview Level 1 urban trauma center, compassionate and culturally sensitive care and to link them to care in their distant tribal communities. The specific aims include 1) interview Native healers to gather information on culture-specific aspects of recovery from traumatic injury and on linking care to tribal communities, 2) conduct a randomized controlled trial to evaluate the implementation and effectiveness of the intervention. The investigators hypothesize that intervention patients will demonstrate greater improvement than controls in post-traumatic stress disorder (PTSD) symptoms, depression, functioning, diagnoses, and fewer new injuries during the 6 months after the index injury.

DETAILED DESCRIPTION:
American Indians are at a greater risk for traumatic life events than the general population and compared to Whites they have a 2.04 (95% CI 1.11, 3.54) fold increased risk of Post Traumatic Stress Disorder (PTSD) symptoms. Among more than 2,900 injured trauma survivors treated at 69 hospitals nationwide, American Indians had the highest risk of all racial/ethnic groups of developing symptoms consistent with a diagnosis of PTSD 12 months after injury. Similarly, among 269 traumatically injured patients hospitalized at 2 level 1 trauma centers in the Western U.S., PTSD and peritraumatic dissociative symptoms were significantly more frequent among American Indians compared to Whites.

Nine percent of 6,000 injured trauma survivors admitted annually to the Harborview Level 1 trauma center are American Indian. Approximately 40 percent of these patients live more than 50 miles from the trauma center, including tribal communities in Eastern Washington and the Olympic Peninsula. Through prior work, researchers have found that care management interventions can reduce PTSD symptoms among diverse injured urban patients. Investigators from the Center of Excellence suggest that American Indian trauma survivors may have unique culture-specific idioms for posttraumatic distress (e.g. "wounded spirit"), and that trauma interventions with indigenous approaches may be productively applied to patients suffering from posttraumatic distress.(5)

In an effort to reduce the risk of PTSD and other general symptoms of trauma among American Indians, we plan to conduct a pilot study to develop and evaluate an American Indian culture specific care management intervention, Staying Connected.

Based on the Trauma Survivors and Support Study (TSOS), the purpose of Staying Connected is to provide American Indian trauma patients, treated at the Harborview Level 1 urban trauma center, compassionate and culturally sensitive care and to link them to care in their distant tribal communities. The specific aims include 1) interview Native healers to gather information on culture-specific aspects of recovery from traumatic injury and on linking care to tribal communities, 2) conduct a randomized controlled trial to evaluate the implementation and effectiveness of the intervention. We hypothesize that intervention patients will demonstrate greater improvement than controls in PTSD symptoms, depression, functioning, diagnoses, and fewer new injuries during the 6 months after the index injury.

ELIGIBILITY:
Inclusion Criteria:

1. Harborview trauma patient 18 years or older
2. self identify as American Indian or Alaska Native
3. speak English

Exclusion Criteria:

1. non-American Indian or Alaska Native status reported
2. monolingual non-English speaking status
3. age < 18 years
4. old head, spinal cord or other injuries that prevent participation in the interview
5. any self-inflicted injury, active psychosis, mania, and victims of intimate partner violence who require immediate intervention
6. currently incarcerated patients or a recent history of severe violence which will likely yield criminal charges

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Post Traumatic Stress Disorder Symptoms assessed by a PCL score | Six months

SECONDARY OUTCOMES:
Depression, Composite International Diagnostic Interview and alcohol abuse/dependence | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Doug Zatzick, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States